CLINICAL TRIAL: NCT01851174
Title: A Phase II Study Evaluating Bi-weekly Dosing of Gemcitabine Plus Nab-Paclitaxel in the First Line Treatment of Surgically Unresectable/Metastatic Pancreatic Cancer
Brief Title: Study to Evaluate Bi-weekly Dosing of Gemcitabine Plus Nab-Paclitaxel to Treat Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Leaving Site
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRMC 12-25
Record Dates: First submitted 2013-02-15; First posted 2013-05-10 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Carcinoma Non-resectable; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine and nab-Paclitaxel (Experimental): Gemcitabine (1,000 mg/m^2) administered intravenously on days 1 and 15, every 28 days
  nab-Paclitaxel (125 mg/m^2) administered intravenously on days 1 and 15, every 28 days
  Interventions: Drug: Gemcitabine; Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Patients will receive Gemcitabine (1,000 mg/m^2) IV over 30 minutes after nab-paclitaxel infusion
  Other Names: Gemzar
Drug: nab-Paclitaxel — Patients will receive nab-Paclitaxel (125 mg/m^2) IV over 30 minutes before Gemcitabine infusion
  Other Names: Abraxane

SUMMARY:
To determine whether the occurrence of adverse events can be decreased by moving to a bi-weekly schedule of gemcitabine plus nab-Pacitaxel for the treatment of unresectable/metastatic pancreatic cancer.

DETAILED DESCRIPTION:
This study will help determine whether the occurrence of adverse events can be decreased by moving to a bi-weekly, opposed to a weekly, dosing schedule of gemcitabine plus nab-Pacitaxel for the treatment of unresectable/metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically-proven unresectable/metastatic pancreatic adenocarcinoma.
2. Patient has one or more radiographically measurable tumor.
3. Patients may have received prior adjuvant chemotherapy or radiation therapy (RT).
4. Age ≥ 18 years.
5. Patient must have read, understood, and provided written informed consent and HIPAA authorization after full explanation of the nature of the study.
6. ECOG performance status 0 - 2 and an expected survival of at least 3 months.
7. Acceptable hematological parameters within 2 weeks of commencing study therapy as follows:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
   * Platelet count ≥ 100 x 10^9/L
   * Hemoglobin (Hgb) ≥ 9g/dl
8. Patients with adequate organ function as measured by:

   A. Cardiac: American Heart Association Class I: Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain.

   B. Hepatic: Bilirubin ≤ 2.0 mg/ and ALT and AST ≤ 1.5x the upper limit of normal.

   C. Renal: Creatinine ≤ 1.5 mg/dl and no other chronic kidney disease.
9. Women must meet one of the following criteria:

   * Post-menopausal for at least one year
   * Surgically incapable of child-bearing
   * Utilizing a reliable form of contraception for the duration of study participation. Women of child-bearing potential must have a negative serum β-HCG within 7 days of study drug administration.

Exclusion Criteria:

1. Previous use of nab-Paclitaxel for treatment of pancreatic cancer either as monotherapy or combination in neo-adjuvant, adjuvant, or the metastatic setting.
2. Previous use of any chemotherapy or radiation therapy for metastatic disease.
3. Patient has known brain metastases, unless previously treated and well-controlled for at least 3 months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart).
4. Other significant active or chronic infection.
5. History of active other malignancy excluding basal or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia.
6. Pregnant or nursing females.
7. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
8. Major surgery, other than diagnostic surgery within 4 weeks of study entry.
9. Patient requires a legal authorized representative for consenting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madappa Kundranda, MD, PhD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Nab-Paclitaxel: Gemcitabine (1,000 mg/m^2) administered intravenously on days 1 and 15, every 28 days
  nab-Paclitaxel (125 mg/m^2) administered intravenously on days 1 and 15, every 28 days
  Gemcitabine: Patients will receive Gemcitabine (1,000 mg/m^2) IV over 30 minutes after nab-paclitaxel infusion
  nab-Paclitaxel: Patients will receive nab-Paclitaxel (125 mg/m^2) IV over 30 minutes before Gemcitabine infusion
Period: Overall Study
Arm/Group | Gemcitabine and Nab-Paclitaxel
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The information required here was not captured. The investigator(s) are no longer at the site and no additional information was left.
Arm/Group | Gemcitabine and Nab-Paclitaxel
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Based on Toxicity Profile of Adverse Events.
Description: Determine the toxicity profile (decrease in hematological and non-hematological treatment-related AE's) with bi-weekly dosing of gemcitabine plus nab-Paclitaxel
Time Frame: One year
Population: The information required here was not captured. The investigator(s) are no longer at the site and no additional information or instruction was left.
Arm/Group | Gemcitabine and Nab-Paclitaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: Progression Free Survival Time
Description: Determine progression free survival time with this regimen
Time Frame: One year
Population: The information required here was not captured. The investigator(s) are no longer at the site and no additional information or instruction was left. Data were not collected
Arm/Group | Gemcitabine and Nab-Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: There is no information available that reflects this information. The information required here was not captured. The investigator(s) are no longer at the site and no additional information or instruction was left.
Description: This information was not recorded and is not available. The investigator(s) are no longer at the site and no additional information or instruction was left.
Arm/Group | Gemcitabine and Nab-Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes